CLINICAL TRIAL: NCT05046314
Title: The Efficacy and Safety of TK216 in Subjects With Relapsed or Refractory Ewing's Sarcoma：a Phase II Clinical Trial in China
Brief Title: A Clinical Study of TK216 in Patients With Relapsed or Refractory Ewing's Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK216-001
Record Dates: First submitted 2021-08-24; First posted 2021-09-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma, Ewing
Keywords: Relapsed and refractory Ewing's Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TK216+Vincristin (Experimental)
  Interventions: Biological: TK216+Vincristin

INTERVENTIONS:
Biological: TK216+Vincristin — TK216 was continuously administered for 14 days，then rest for 14 days. Vincristin is given before TK216 only in the first day of each cycle, the first cycle of VCR is 0.75mg/m^2 and 1.5mg/m^2 from the second cycle，every 28 days is a study cycle.

SUMMARY:
This study is a multicenter, single-arm, open-label Phase II clinical trial evaluating TK216 in combination with vincristine in the treatment of relapsed or refractory Ewing sarcoma (ES) including Ewing's sarcoma family tumors (ESFTs).

DETAILED DESCRIPTION:
Ewing sarcoma is characterized by genomic rearrangements resulting in over-expression of ets family transcription factors driving tumor progression. TK216 is designed to inhibit this effect by inhibiting downstream effects of the EWS-FLI1 transcription factor. Based on USA RP2D result, designed as a single arm, multicenter open-label study，this study is the first study of TK216 in Chinese subjects with Ewing sarcoma. The study is designed to establish safety and efficacy data in combination with vincristine to assess the potential of TK216 for further development.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for this study:

1. Willing to sign the informed consent form.
2. Participants with relapsed or refractory ES (including ESFT, except Ewing-like sarcoma) confirmed by cytohistology or molecular biology.
3. Life expectancy of at least 3 months.
4. Participants age ≥ 14 years, regardless of gender.
5. At least one measurable lesion according to RECIST version 1.1.
6. Agree to have a central venous catheter in place prior to initiating infusion of study drug.
7. Prior radiotherapy is allowed if ≥ 2 weeks must have elapsed for local palliative external beam radiotherapy; ≥ 6 months must have elapsed if systemic radiotherapy, external craniospinal irradiation or > 50% pelvic radiotherapy; and ≥ 6 weeks must have elapsed for other substantial bone marrow radiotherapy before the first dose. Participants who have received brain radiotherapy must have completed whole brain radiotherapy and/or gamma knife surgery at least 4 weeks prior to enrollment.
8. Stem Cell Transplant or Rescue without TBI：no evidence of active graft-versus-host disease and ≥ 3 months must have elapsed since transplant.
9. Symptomatic CNS metastases must have been treated and remain stable for at least 4 weeks prior to the first dose of the study drug, or patients with asymptomatic brain metastases.
10. Adequate hematological and organ functions fulfilling the following laboratory requirements, and these results should be obtained within 7 days prior to the first dose:
11. ECOG performance score 0-2.
12. Cardiac ejection fraction ≥ 50% or shortening fraction ≥ 28%.
13. Eligible male and female participants of childbearing potential must consent to use reliable methods of contraception with their partners for at least 4 weeks before the start of protocol therapy, for the duration of study participation, and for at least 6 months after the last dose. Women of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose.
14. Without any contraindication to vincristine.

Exclusion Criteria:

Participants will not be enrolled if they meet any of the following exclusion criteria:

1. Current participation in another therapeutic clinical trial.
2. Having received anti-tumor chemotherapy, targeted therapy or immunotherapy within 4 weeks prior to the first dose; having received Chinese herbal medicine or Chinese patent medicine-based therapies with definite anti-tumor indications within 3 weeks before study drug usage.
3. Having received systemic corticosteroids or other systemic immunosuppressive agents within 14 days prior to study, with the following exceptions:

   1. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption;
   2. Short-term (≤ 7 days), prophylactic use of corticosteroids or for the treatment of non-autoimmune diseases
4. Unresolved, > Grade 1 toxicity related to prior anti-tumor therapy prior to the study, according to the CTCAE version 5.0.
5. History of previous cancer, except squamous cell or basal -cell carcinoma of the skin or any in situ carcinoma that has been completely resected, which required therapy within the previous 3 years.
6. Any of the following within 6 months: uncontrolled congestive heart failure (NYHA III-IV); uncontrolled angina; onset of cerebrovascular event or transient ischemic attack; pulmonary embolism; deep vein thrombosis and symptomatic bradycardia that require the use of antiarrhythmic drugs.
7. History of QTc prolongation
8. History of additional risk factors for torsades de pointes
9. Use of concomitant medications that may increase or possibly increase the risk to prolong the QTc interval and/or induce torsades de pointes ventricular arrhythmia.
10. Having received surgical therapies (except diagnostic surgery, such as tumor biopsy, diagnostic puncture, etc.), including surgical and interventional therapies, within 4 weeks prior to treatment.
11. Systemic use of antibiotics for ≥ 7 days within 4 weeks before TK216 treatment, or have fever of unknown origin (> 38.5 °C）
12. Positive test results for hepatitis B surface antigen, hepatitis C antibody and HIV antibody during screening.
13. Females who are pregnant or lactating.
14. Have taken potent inducers or inhibitors of CYP3A4, potent inhibitors of CYP2C19 within 2 weeks prior to the first dose of study drug, or substrates of CYP3A4/CPY2C19 with a narrow therapeutic window.
15. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or study drug management, or may interfere with the interpretation of the study results.
16. Participants who are not suitable for participating in this study due to any reason as judged by the investigator.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-09-13 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (IRC) | Up to 2 years after TK216 introduction
  Determination of the Objective Response Rate of all patients by IRC

SECONDARY OUTCOMES:
Objective Response Rate (Investigator) | Up to 2 years after TK216 introduction
  Determination of the Objective Response Rate of all patients by investigators
Progression-free survival (PFS) | Up to 2 years after TK216 introduction
  Determination of the progression-free survival of all patients
Overall survival (OS) | Up to 2 years after TK216 introduction
  Determination of the overall survival times of all patients
Disease control rate (DCR) | Up to 2 years after TK216 introduction
  Determination of the disease control rate of all patients
Duration of remission (DOR) | Up to 2 years after TK216 introduction
  Determination of the duration of remission of all patients
Drug concentration in plasma | Up to 2 years after TK216 introduction
  Determination of drug concentration in plasma of all patients
Number of patients with adverse events | Up to 2 years after TK216 introduction
  Adverse event type, incidence, duration, correlation with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yao, Principal Investigator — Shanghai 6th People's Hospital
Locations (8):
- China (8):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institude & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang